CLINICAL TRIAL: NCT04487119
Title: Pediatric COVID-19 Infection; Do Clinical Features and Hematological Parameters Predict the Need for ICU Admission?
Brief Title: Hematology and Clinical Picture in Pediatric COVID-19 Infection
Status: Completed | Type: Observational
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Shaimaa Reda Abdelmaksoud, MD Lecturer pediatrics, Benha University
Other Study IDs: RC 6-7-2020
Record Dates: First submitted 2020-07-24; First posted 2020-07-27 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Covid19
Keywords: COVID19; hematology; pediatric
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is to discuss the different clinical presentations, hematological and laboratory abnormalities in pediatric COVID-19 infection.

DETAILED DESCRIPTION:
This retrospective observational study will be conducted at Benha University Hospital, Benha, Egypt; after approval by the local ethical committee of Faculty of Medicine, Benha University, Egypt.

We will include in this retrospective study all pediatric patients who were admitted with confirmed COVID-19 infection with age range from birth to 18 years during the period from April 2020 till July 2020. The diagnosis of COVID-19 infection is based on positive SARS-CoV-2 RNA detection in throat swab specimens by PCR.

All data including demography information, contact history, previous history, clinical symptoms, clinical examination on admission, and hematology and laboratory information will be obtained from inpatient medical records.

ELIGIBILITY:
Inclusion Criteria:

-inpatient confirmed COVID-19 infection by PCR

Exclusion Criteria:

* patients with records missing hematology and/or laboratory data,
* patients transfered to other medical facilities with unknown outcomes,
* patients with age older than 18 years from the study.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: all pediatric patients who were admitted with confirmed COVID-19 infection with age range from birth to 18 years during the period from April 2020 till July 2020. The diagnosis of COVID-19 infection is based on positive SARS-CoV-2 RNA detection in throat swab specimens by PCR.
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2020-08-12 (Actual); Primary Completion 2020-08-20 (Actual); Study Completion 2020-08-23 (Actual)

PRIMARY OUTCOMES:
hematological findings | at time of admission
  hematological indices; TLC, absolute lymphocytic count, absolute neutrophil count platelet count, N/L ratio and CRP in pediatric COVID-19 infection

SECONDARY OUTCOMES:
clinical presentations | at time of admission
  proportion of patients with respiratory and GIT symptoms, proportion of patients needs ICU admission relation between severity and hematologic indices

CONTACTS AND LOCATIONS:
Overall Officials: Shaimaa R Abdelmaksoud, MD, Principal Investigator — Benha University; Rana A Khashaba, MD, Study Chair — Benha University; Effat H Assar, MD, Study Chair — Benha University; Rasha S Eldesouky, MD, Study Chair — Benha University
Locations (1):
- Benha Faculty of Medicine, Banhā, Qalyubia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang D, Hu B, Hu C, Zhu F, Liu X, Zhang J, Wang B, Xiang H, Cheng Z, Xiong Y, Zhao Y, Li Y, Wang X, Peng Z. Clinical Characteristics of 138 Hospitalized Patients With 2019 Novel Coronavirus-Infected Pneumonia in Wuhan, China. JAMA. 2020 Mar 17;323(11):1061-1069. doi: 10.1001/jama.2020.1585. PMID 32031570
- [Background] Fan BE, Chong VCL, Chan SSW, Lim GH, Lim KGE, Tan GB, Mucheli SS, Kuperan P, Ong KH. Hematologic parameters in patients with COVID-19 infection. Am J Hematol. 2020 Jun;95(6):E131-E134. doi: 10.1002/ajh.25774. Epub 2020 Mar 19. No abstract available. PMID 32129508